CLINICAL TRIAL: NCT00612664
Title: A Randomized, Multi-Dose, Open-Label, Phase II Study of BMS-663513 as a Second-Line Monotherapy in Subjects With Previously Treated Unresectable Stage III or IV Melanoma
Brief Title: Phase II, 2nd Line Melanoma - RAND Monotherapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CA186-006
Record Dates: First submitted 2008-01-30; First posted 2008-02-12 (Estimated); Last update posted 2015-10-12 (Estimated); Status verified 2015-09

CONDITIONS: Melanoma
MeSH Terms: conditions — Melanoma | interventions — urelumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Arm 1 (Active Comparator): 0.1 mg/kg every 3 weeks
  Interventions: Drug: Anti-CD137 (4-1BB) (BMS-663513)
- Arm 2 (Active Comparator): 1 mg/kg every 3 weeks
  Interventions: Drug: Anti-CD137 (4-1BB) (BMS-663513)
- Arm 3 (Active Comparator): 1 mg/kg every 6 weeks
  Interventions: Drug: Anti-CD137 (4-1BB) (BMS-663513)
- Arm 4 (Active Comparator): 5 mg/kg every 3 weeks
  Interventions: Drug: Anti-CD137 (4-1BB) (BMS-663513)

INTERVENTIONS:
Drug: Anti-CD137 (4-1BB) (BMS-663513) — IV solution, IV, until PD or toxicity

SUMMARY:
The main purpose of this study is to estimate the proportion of patients with a type of skin cancer called melanoma who are progression free, (that is, the cancer has not gotten substantially worse), when treated with Anti-CD137 (4-1BB) (BMS-663513) at 0.1 mg/kg, 1 mg/kg or 5 mg/kg every 3 weeks or 1 mg/kg every 6 weeks

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have been previously treated with one line of systemic anti-cancer therapy (non-experimental or experimental) for metastatic disease, and relapsed, failed to respond (CR or PR) or did not tolerate that regimen. If the treatment has been administered as an adjuvant and/or neoadjuvant therapy, the subject must have documented disease progression from the last treatment and also received one additional line of systemic therapy for metastatic disease.
* Men and women, who are at least 18 years of age

Exclusion Criteria:

* Ocular or mucosal melanoma
* Complete surgical resection of all identifiable sites of disease
* Symptomatic brain metastasis. Subjects with signs or symptoms suggestive of brain metastasis are not eligible unless brain metastases are ruled out by computerized axial tomography (CT) scan or magnetic resonance imaging (MRI). Subjects with stable brain metastasis and those who were previously treated with radiotherapy or surgery must have no current evidence of symptomatic brain metastasis and are off steroid therapy for at least 4 weeks prior to randomization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 158 (Actual)
Dates: Start 2008-03; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Radiographic imaging, photographic and clinical evaluation will be used for tumor assessment to determine 6-month progression-free survival rate | every 6 weeks starting at week 12 after randomization

SECONDARY OUTCOMES:
Safety profiles | throughout the study
Disease response rate | end of study
Disease control rate | end of study
1-year survival | end of study
Pharmacokinetics | throughout the study
Pharmacodynamics | throughout the study
Biomarkers | throughout the study

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (31):
- United States (10):
  - The Angeles Clinic & Research Institute, Los Angeles, California
  - Yale University School Of Medicine, New Haven, Connecticut
  - Oncology Specialists, S.C., Park Ridge, Illinois
  - Indiana University Melvin And Bren Simon Cancer Center, Indianapolis, Indiana
  - Harry & Jeanette Weinberg Cancer Inst At Franklin Square, Baltimore, Maryland
  - Dana-Farber Cancer Inst, Boston, Massachusetts
  - Mem Sloan-Ket Can Ctr, New York, New York
  - Blumenthal Cancer Center, Carolinas Medical Center, Charlotte, North Carolina
  - Providence Portland Medical Center, Portland, Oregon
  - University Of Texas, Houston, Texas
- Canada (3):
  - Local Institution, Calgary, Alberta
  - Local Institution, Edmonton, Alberta
  - Local Institution, Montreal, Quebec
- Denmark (2):
  - Local Institution, Aarhus C
  - Local Institution, Odense C
- France (4):
  - Local Institution, Lille
  - Local Institution, Paris
  - Local Institution, Vandœuvre-lès-Nancy
  - Local Institution, Villejuif
- Germany (7):
  - Local Institution, Homburg / Saar
  - Local Institution, Jena
  - Local Institution, Kiel
  - Local Institution, Mainz
  - Local Institution, Mannheim
  - Local Institution, Tübingen
  - Local Institution, Würzburg
- Italy (5):
  - Local Institution, Genove
  - Local Institution, Milan
  - Local Institution, Napoli
  - Local Institution, Padua
  - Local Institution, Siena

REFERENCES:
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx